CLINICAL TRIAL: NCT05312632
Title: A Multi-center, Open-label Phase 4 Study Evaluating the Efficacy and Safety of Safinamide Mesilate as Add-on Therapy to Levodopa in Parkinson's Disease Patients With Motor Fluctuation in South Korea
Brief Title: A Study to Evaluate the Efficacy and Safety of Safinamide Mesilate as Add-on Therapy to Levodopa in Parkinson's Disease Participants With Motor Fluctuation in South Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME2125-M082-401
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safinamide Mesilate (Experimental): Participants with parkinson's disease will be administered Safinamide Mesilate 50 milligram (mg) tablet, orally, once daily as add-on therapy to levodopa for up to 2 weeks. After 2 weeks, at the discretion of an investigator, dose of Safinamide Mesilate will be increased to 100 mg tablets (two tablets of 50 mg each), orally, once daily for up to 18 weeks.
  Interventions: Drug: Safinamide Mesilate

INTERVENTIONS:
Drug: Safinamide Mesilate — Safinamide Mesilate oral tablets.
  Other Names: Equfina; ME2125

SUMMARY:
The primary purpose of this study is to evaluate the change at the 18th week from baseline in daily "off" time measured by participant diary and Parkinson's Disease Questionnaire-39 (PDQ-39) in participants with Parkinson's Disease who are receiving levodopa.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age greater than or equal to (>=) 19 years at the time of informed consent
2. Participants who meet the clinical diagnostic criteria of Movement Disorder Society (MDS) diagnostic criteria 2015 for Parkinson's disease, have motor fluctuations with >=1.5 hours of "off" time throughout the day which is confirmed at the time of Screening, and take levodopa 3 or more times a day
3. Parkinson's Disease participants who are receiving levodopa without Catechol O-methyltransferase (COMT) inhibitor and/or Monoamine oxidase-B (MAO-B) inhibitor
4. Be able to maintain an accurate and complete diary with the help of a caregiver as needed, recording "on" time, "on" time with dyskinesia, "off" time, and time asleep
5. Be able to provide written informed consent
6. Participants whose cognitive function, at the discretion of an investigator, is at a level appropriate to participate in the clinical trial (that is., with a Global Deterioration Scale [GDS] score of 3 or less or a Clinical Dementia Rating [CDR] of 0.5 or less within 3 months prior to screening)

Exclusion Criteria:

1. Females who are planning for pregnancy, pregnant or breastfeeding
2. Prior use of safinamide
3. If participants have previously taken medication such as COMT inhibitor and/or MAO-B inhibitor, they have to take appropriate wash-out period for each medication (3 days for COMT inhibitor; 14 days for MAO-B inhibitor)
4. Use of medications for depression or psychosis within 5 weeks prior to screening
5. History of allergic response to levodopa, or other anti-Parkinsonian agents
6. Hypersensitivity or contraindications to MAO-B inhibitors
7. Confirmed ophthalmologic history including any of the following conditions: albino participants, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (that is, 20/70 on Snellen Chart), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or diabetic retinopathy
8. Participants who did not consent to having at least 7 days of washout period prior to visit 2, if known to take narcotic analgesics 7 days prior to screening visit (example, pethidine hydrochloride-containing products, tramadol hydrochloride, or tapentadol hydrochloride)
9. History of serotonergic medications administration (example, tricyclic antidepressants, tetracyclic antidepressants, selective serotonin reuptake inhibitors, serotonin-noradrenaline reuptake inhibitors, selective noradrenaline reuptake inhibitor, or noradrenergic and serotonergic antidepressant) within 5 weeks prior to screening visit
10. Administering central nervous system stimulants (example, methylphenidate hydrochloride, lisdexamfetamine mesilate)
11. Administering dextromethorphan
12. Participants with clinically significant liver function abnormalities defined as greater than (>) 1.5 times of the upper limit of the normal range of total bilirubin or >3 times of the upper limit of the normal range of Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST); re-examination and re-screening are allowed once within the screening period
13. Have a history of hypersensitivity to any of the ingredients of the product
14. Currently enrolled in another clinical trial or used any investigational drug/biologics or device within 30 days or 5*the half-life, whichever is longer, preceding informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- South Korea (20):
  - Eisai Site #11, Busan
  - Eisai Site #20, Busan
  - Eisai Site #3, Busan
  - Eisai Site #16, Daegu
  - Eisai Site #2, Daegu
  - Eisai Site #19, Daejeon
  - Eisai Site #10, Gwangju
  - Eisai Site #12, Gyeonggi-do
  - Eisai Site #15, Gyeonggi-do
  - Eisai Site #17, Gyeonggi-do
  - Eisai Site #5, Gyeonggi-do
  - Eisai Site #14, Incheon
  - Eisai Site #13, Seoul
  - Eisai Site #18, Seoul
  - Eisai Site #1, Seoul
  - Eisai Site #4, Seoul
  - Eisai Site #6, Seoul
  - Eisai Site #7, Seoul
  - Eisai Site #8, Seoul
  - Eisai Site #9, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Oh E, Cheon SM, Cho JW, Sung YH, Kim JS, Shin HW, Kim JM, Park MY, Kwon DY, Ma H 2nd, Park JH, Koh SB, Choi SM, Park J, Lee PH, Ahn TB, Kim SJ, Lyoo CH, Lee HW, Kim J, Lee Y, Baik JS. Efficacy and safety of safinamide in Parkinson's disease patients with motor fluctuations without levodopa dosage escalation over 18 weeks: KEEP study. J Neural Transm (Vienna). 2025 Mar;132(3):431-441. doi: 10.1007/s00702-024-02851-6. Epub 2024 Nov 14. PMID 39540934

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 20 investigative sites in South Korea from 05 April 2022 to 25 May 2023.
Pre-assignment Details: A total of 222 participants were screened, of which 21 were screen failures and 201 were enrolled and treated in this study.
Groups:
- Safinamide Mesilate 100 mg: Participants with parkinson's disease received safinamide mesilate 50 milligram (mg) tablet, orally, once daily as add-on therapy to levodopa for up to 2 weeks. After 2 weeks, at the discretion of an investigator, dose of safinamide mesilate was increased to 100 mg (two tablets of 50 mg each), orally, once daily for up to 18 weeks.
Period: Overall Study
Arm/Group | Safinamide Mesilate 100 mg
Started | 201
Safety Analysis Population | 199
Full Analysis Population | 196
Completed | 162
Not Completed | 39
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 10
Not completed — Lack of Efficacy | 4
Not completed — Non-compliance with study procedures | 9
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: The safety analysis population included participants who received at least 1 dose of study drug and completed at least 1 post-dose safety assessment.
Groups:
- Safinamide Mesilate 100 mg: Participants with parkinson's disease received safinamide mesilate 50 mg tablet, orally, once daily as add-on therapy to levodopa for up to 2 weeks. After 2 weeks, at the discretion of an investigator, dose of safinamide mesilate was increased to 100 mg (two tablets of 50 mg each), orally, once daily for up to 18 weeks.
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 95
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 199

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Daily "OFF" Time at Week 18
Description: Participants received diary card and information on daily 'off' time and 'on' time was collected. At 30-minutes intervals throughout the period, the participant/caregiver recorded whether the participant was in an "on" phase, in an "on" phase with dyskinesia, in an "off" phase, or asleep. An "off" phase was defined as lack of mobility, bradykinesia, or akinesia whereas in an "on" phase, the participant functioned as well as can be expected for that participant, irrespective of whether or not he or she is having dyskinesia. The daily "off" time was defined as the mean of the total daily "off" time during the last two 24 hours dairy recording periods.
Time Frame: Baseline, Week 18
Population: The full analysis set (FAS) included participants who received at least 1 dose of study drug and had at least 1 record of daily "off" time or the Parkinson's disease questionnaire (PDQ-39) after dosing. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 189
hours | -0.8 [-11.2 to 3.7]
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p < 0.001, Wilcoxon signed rank test

2. Primary Outcome: Change From Baseline in PDQ-39 Score at Week 18
Description: The PDQ-39 was a self-reported outcome or rater-reported outcome of 39 questions relating to 8 domains: mobility (Questions 1-10), activities of daily living (ADL) (Questions 11-16), emotional well-being (Questions 17-22), stigma (Questions 23-26), social support (Questions 27-30), cognition (Questions 31-33), communication (Questions 34-36) and bodily discomfort (Questions 37-39). Each question was answered on a 5-point scale from 0 (Never) to 4 (Always/Cannot Do At All). Scores were calculated by summing the answers to the questions in the domain and converting to a total score scale from 0 to 100. Higher scores were associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 18
Population: The FAS included all participants who received at least 1 dose of study drug and had at least 1 record of daily "off" time or PDQ-39 after dosing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 196
score on a scale | -2.7 (10.3)
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p < 0.001, Wilcoxon signed rank test

3. Secondary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating (MDS-UPDRS) Part 3 at Week 18
Description: MDS-UPDRS rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts: Part 1: Non-motor aspects of experiences of daily living; Part 2: Motor aspects of experiences of daily living; Part 3: Motor examination; Part 4: Motor complications. Part 3 section of scale consisted of 18 items, with 33 separate ratings being performed on scale from 0 (normal) to 4 (severe). The total score ranged from 0 to 132, with a lower score=better motor function; higher score=more severe motor symptoms.
Time Frame: Baseline, Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 196
score on a scale | -1.7 (8.4)
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p < 0.001, Wilcoxon signed rank test

4. Secondary Outcome: Change From Baseline in MDS-UPDRS Part 4 at Week 18
Description: The MDS-UPDRS rating tool was used to follow longitudinal course of Parkinson's Disease. It was made up of 4 parts that assess: Part 1: Non-motor aspects of experiences of daily living; Part 2: Motor aspects of experiences of daily living; Part 3: Motor examination; Part 4: Motor complications. Part 4 raters use historical/objective information to assess 2 motor complications, dyskinesias and motor fluctuations including OFF-state dystonia. Raters use information from participant, caregiver, and the examination to answer 6 questions. The duration of disability caused and functional impact of any dyskinesias experienced by the participant were rated on a scale of 0 to 4. 6 items being performed on scale from 0 (normal) to 4 (severe), where the total score ranged from 0 to 24, lower score indicated better motor function and higher score indicated more severe motor symptoms.
Time Frame: Baseline, Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 196
score on a scale | -0.7 (2.1)
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p < 0.001, Wilcoxon signed rank test

5. Secondary Outcome: Change From Baseline in King's Parkinson's Disease Pain Scale (KPPS) at Week 18
Description: KPPS is a Parkinson's Disease-specific pain scale that evaluated the localization, frequency, and intensity of pain. It has 14 items in 7 domains: 1. Musculoskeletal pain; 2. Chronic pain; 3. Fluctuation-related pain; 4. Nocturnal pain; 5. Oro-facial pain; 6. Discoloration, Oedema/Swelling pain; 7. Radicular pain. Each item was scored by severity (0 [none] to 3 [very severe]) multiplied by frequency (0 [never] to 4 [all the time]), resulting in a subscore of 0 to 12, the sum of which gives the total score which ranged from 0 to 168. Higher scores indicated more severity and frequency of pain.
Time Frame: Baseline, Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 196
score on a scale | -1.5 (11.3)
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p = 0.013, Wilcoxon signed rank test

6. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) at Week 18
Description: The MMSE is a brief practical screening test for cognitive dysfunction. The test consists of 5 sections (orientation, registration, attention and calculation, recall, and language) and has a total possible score of 30. Total scores ranged from 0 (most impaired) to 30 (no impairment). MMSE used to assess the severity of cognitive dysfunction, with a higher score indicating better cognitive state.
Time Frame: Baseline, Week 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 196
score on a scale | 0.2 (1.7)
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p = 0.053, Wilcoxon signed rank test

7. Secondary Outcome: Change From Baseline in Daily "ON" Time Without Dyskinesia at Week 18
Description: Participants received diary card and information on daily 'off' time and 'on' time was collected. At 30-minute intervals throughout the period, the participant/caregiver recorded whether the participant was in an "on" phase, in an "off" phase, or asleep. An "off" phase was defined as lack of mobility, bradykinesia, or akinesia whereas in an "on" phase, the participant functioned as well as can be expected for that participant, irrespective of whether or not he or she is having dyskinesia. The daily "on" time was defined as the sum of the time without dyskinesia during the on phase to number of days completed in the diary.
Time Frame: Baseline, Week 18
Population: The FAS included all participants who received at least 1 dose of study drug and had at least 1 record of daily "off" time or PDQ-39 after dosing. Here, Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 189
hours | 0.7 [-6.2 to 10.0]
Statistical Analysis 1: Comparison: Safinamide Mesilate 100 mg; Test type: Other; p < 0.001, Wilcoxon signed rank test

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE was defined as an adverse event (AE) that emerges during treatment, having been absent at pretreatment (Baseline) or reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or worsens in severity during treatment relative to the pretreatment state, when the AE is continuous. SAE was any untoward medical occurrence that at any dose: results in death, was life-threatening, inpatient hospitalization, requires prolongation of existing hospitalization, results in persistent or significant disability/incapacity, was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug), was a medically significant event.
Time Frame: From the first dose of the study drug up to end of the treatment (up to Week 18)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Safinamide Mesilate 100 mg
Number analyzed (Participants) | 199
Participants
  TEAEs | 80
  SAEs | 4

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug up to end of the treatment (up to Week 18)
Description: The safety analysis population included participants who received at least 1 dose of study drug and completed at least 1 post-dose safety assessment.
Arm/Group | Safinamide Mesilate 100 mg
All-Cause Mortality (participants affected / at risk) | 0/199
Serious Adverse Events (participants affected / at risk) | 4/199
Other Adverse Events (participants affected / at risk) | 56/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safinamide Mesilate 100 mg (N=199)
Cartilage injury (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Condition aggravated (General disorders) | 1
COVID-19 (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safinamide Mesilate 100 mg (N=199)
Dyskinesia (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 3
Dystonia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Overdose (Injury, poisoning and procedural complications) | 13
Nausea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
COVID-19 (Infections and infestations) | 5
Drug ineffective (General disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 4
Delusion (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT05312632/Prot_SAP_000.pdf